CLINICAL TRIAL: NCT06150833
Title: Efficacy, Safety and Pharmacokinetics of Boya Intravenous Immunoglobulin (IVIG) in Participants With Primary Immunodeficiency
Brief Title: Efficacy and Safety and Pharmacokinetics of Boya IVIG
Acronym: Boya
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Boya Bio Pharmaceutical Group Co Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BoyaIVIG
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Primary Immunodeficiency Disease
Keywords: BOYA; IVIG; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Patients with primary immunodeficiency will switch to Boya IVIG and optimize the posology in a run-in period of 2 to 6 administrations. In the one-year test period, the patients will receive the test IVIG at 21- or 28-day intervals and be followed. IgG trough levels will be collected from all participants, at all visits. The remaining pharmacokinetic parameters will be measured between visits 4 and 5 in 20 adult participants, collecting additional blood samples.
Masking Description: The trial will be open-label and single-arm. Therefore, there will be no randomization or blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Boya IVIG (Experimental): Patients with primary immunodeficiency will switch to Boya IVIG and optimize the posology in a run-in period of 2 to 6 administrations. In the one-year test period, the patients will receive the test IVIG at 21- or 28-day intervals and be followed. The minimum IgG concentration will be measured in all participants at all visits. The other pharmacokinetic parameters will be measured between visits 4 and 5 in 20 adult participants by taking additional blood samples. An independent Safety Data Monitoring Committee (SDMC) will periodically monitor adverse events.
  Interventions: Biological: Boya IVIG

INTERVENTIONS:
Biological: Boya IVIG — The initial dose and other dose changes will be determined by the investigator on a case-by-case basis aiming to prevent infection and minimum serum IgG levels of 5 g/L. The total number of doses administered will depend on the treatment regimen and run-in period:
  * Between 16 and 20 intravenous injections for participants receiving infusions every 28 days, or;
  * Between 21 and 25 intravenous injections for participants receiving infusions every 21 days
  Other Names: IVIG; BOYA

SUMMARY:
To evaluate the safety, efficacy and pharmacokinetic properties of Boya's IVIG preparation in participants with PID aged less than 60 years and more than 6 years.

DETAILED DESCRIPTION:
This is a phase 3, open-label, prospective, single-group, multicenter study to evaluate the efficacy of IVIG in keeping the average number of serious bacterial infections to less than one per year. The safety and pharmacokinetics (PK) of the investigational product will also be assessed. Fifty male or female participants aged up to 60 years will be selected, with at least 20 participants aged between 06 and 17 years. During the study, at least 20 adult participants will be invited to make up the subgroups evaluating the pharmacokinetic parameters.

The main benefit of IVIG is to help the immune system respond to a wide range of infections, which are often correlated with high morbidity and mortality rates in individuals with PID, particularly in cases of CVID and XLA. In addition, a reduction in the use of medication and hospitalizations is expected, promoting an improvement in the quality of life of these patients.

IVIG therapy is generally safe, although unwanted effects are reported in a proportion ranging from 1% to 81% of patients or infusions, with an average incidence of 30% to 40% among patients and 5% to 15% among infusions. These effects can manifest themselves in varying degrees of intensity, ranging from mild to severe. They can occur immediately, during or shortly after the infusion, as well as late, appearing hours or even days after the procedure. Most adverse events are mild and immediate, occurring in the first few infusions, related to the infusion rate and quickly reversible.

Headache, fever, general malaise, flu-like symptoms, nausea, chills, fatigue, myalgia, low back pain, tachycardia, changes in blood pressure and erythroderma are the most common events. Serious reactions occur in less than 1% of applications and usually with the use of higher doses, indicated in autoimmune and inflammatory diseases.

Special care is needed in patients with comorbidities such as heart disease, nephropathy, liver disease, coagulation disorders (thrombophilia) and diabetes mellitus. In these patients, certain characteristics of IVIG should be assessed, such as the presence of sugars, osmolality, sodium, among others.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of written informed consent.
2. Men or women.
3. Age ≤ 60 years.
4. Diagnosis of PID disease (PID) with a reduction in antibody production due to:

   1. Common variable immunodeficiency (CVID) as defined ESID/PAGID, OR
   2. X-linked agammaglobulinemia (XLA) as defined by ESID/PAGID.
5. Receiving intravenous immunoglobulin replacement therapy at 21- or 28-day intervals at 300 to 600 mg/kg/month for a minimum of 2 months prior to study entry.
6. Absence of episodes of serious bacterial infections with prior use of IV immunoglobulin for at least 3 months prior to screening.
7. Negative pregnancy test (in female participants of childbearing potential); readiness to use reliable contraceptive methods throughout the study period.
8. Patients who have participated in a clinical study with another investigational IVIG may be included if they have a potential benefit in accordance with CNS Res. 251/1997.
9. Participants undergoing treatment with any subcutaneous or intramuscular immunoglobulin may be included by switching to IVIG therapy at the discretion of the investigator, considering the possible benefit to the participant.

Exclusion Criteria:

1. Known intolerance or hypersensitivity to immunoglobulins or components of the test article;
2. Any contraindications to the use of immunoglobulins;
3. Secondary immunodeficiency or conditions potentially causing secondary immunodeficiency such as chronic lymphoid leukemia, lymphoma, multiple myeloma, protein-losing enteropathies or nephropathies, and hypoalbuminemia;
4. Clinically relevant changes in the safety exams are defined as:

   * Blood count

     * Hb < 10.5 g/dL
     * Leukocytes < 3,000 / mm3 or >10,000 cells / mm3
     * Absolute neutrophil count < 1,000 cells/mm3;
   * Coagulation

     * TP and aPTT > 2.5 x ULN
   * Biochemistry

     * glycated hemoglobin > 6.5%
     * total bilirubin and fractions, alkaline phosphatase, ALT, AST, GGT > 2.5 x ULN
     * creatinine above 3mg/dl or creatinine clearance < 30mL/min
   * Urine I.

     * Leukocyturia > 10,000 cells/mL
5. Any cancer either active or resolved within the last 12 months before screening;
6. Receiving any blood products (except intravenous immunoglobulins) during the last 3 months before screening;
7. Any febrile illness within 14 days before enrollment; Note: The patient may be rescreened after recovery.
8. History of thrombotic events (including myocardial infarction, stroke, pulmonary embolism, and deep vein thrombosis) within 6 months before enrollment;
9. Previous use of live attenuated virus vaccines;
10. Selective deficiency of immunoglobulin A (IgA) or known antibodies to IgA;
11. Known drug or alcohol abuse;
12. The need to use other investigational drugs, systemic immunosuppressants, and any other immunoglobulins;
13. Pregnancy or lactation;
14. Inability to comply with the protocol activities;
15. PIDs other than CVID or X-linked agammaglobulinemia
16. Patients infected with HIV, HBV or HCV
17. Patients with AIDS, cystic fibrosis, or active hepatitis B or C.
18. Any other condition that, in the Investigator's opinion may increase the risk of participation in this study.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective (average of acute serious bacterial infections) | Between Visit 0 and Final Visit (through study completion, an average of 1 year)
  The incidence of serious bacterial infections (septicemia, meningitis, visceral abscess, osteomyelitis, and pneumonia) within the 1-year follow-up is less than 1.0 per patient/year in the average of the population.

SECONDARY OUTCOMES:
Assessment of the rate of non-serious infections within one year | Average incidence of non-serious infections per patient between Visit 0 and Final Visit (through study completion, an average of 1 year), as documented as treatment emergent adverse events (TEAEs).
  The incidence of all acute infections except the serious acute bacterial infections within the 1-year follow-up (simple descriptive statistics).
Length of infections | Average number of days for treating infections per patient between visit 0 and final visit (through study completion, an average of 1 year), as documented as treatment emergent adverse events (TEAEs)
  Assessment of the duration of treatment for infections per year
Missing time from school/work | Average number of days off from school/work per patient/month, as documented in the patient's diary (through study completion, an average of 1 year)
  Assessment of time lost at school/work due to infections per month
Hospitalization episodes | Number of days hospitalized per month overall and due to infection, as documented as treatment emergent adverse events - TEAEs (through study completion, an average of 1 year)
  Assessment of hospitalization episodes and length

OTHER OUTCOMES:
Secondary Pharmacokinetic (PK) Objectives | 9 months
  To assess the total IgG serum concentration before each infusion (IgG trough levels), between Visit 4 and Final Visit (through study completion).
Secondary Pharmacokinetic (PK) Objectives | 28 days
  To assess total serum IgG profile (concentration vs time) at specific times between the 5th and 6th infusion
IgG half-life | 28 days
  Determine IgG half-life from concentration vs time curve
Area under the IgG curve | 28 days
  Determine IgG AUC from concentration vs time curve
IgG distribution volume | 28 days
  Determine IgG Vd from concentration vs time curve
IgG elimination constant | 28 days
  Determine IgG Kel from concentration vs time curve
Incidence, severity, and causality of adverse events | 1, 24, and 72 hours after each infusion (through study completion, an average of 1 year)
  Assessment of infusion-related adverse events
Secondary Safety Objective | Incidence, severity, and causality of all treatment-emergent adverse events, except those infusion-related (through study completion, an average of 1 year).
  Assessment of treatment emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Ferrara, Study Director — Azidus Brasil

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.

REFERENCES:
- [Background] Goudouris ES, Rego Silva AM, Ouricuri AL, Grumach AS, Condino-Neto A, Costa-Carvalho BT, Prando CC, Kokron CM, Vasconcelos DM, Tavares FS, Silva Segundo GR, Barreto IC, Dorna MB, Barros MA, Forte WCN. II Brazilian Consensus on the use of human immunoglobulin in patients with primary immunodeficiencies. Einstein (Sao Paulo). 2017;15(1):1-16. doi: 10.1590/S1679-45082017AE3844. PMID 28444082
- [Background] Cordero E, Goycochea-Valdivia W, Mendez-Echevarria A, Allende LM, Alsina L, Bravo Garcia-Morato M, Gil-Herrera J, Gudiol C, Len-Abad O, Lopez-Medrano F, Moreno-Perez D, Munoz P, Olbrich P, Sanchez-Ramon S, Soler-Palacin P, Aguilera Cros C, Arostegui JI, Badell Serra I, Carbone J, Fortun J, Gonzalez-Granado LI, Lopez-Granados E, Lucena JM, Parody R, Ramakers J, Regueiro JR, Riviere JG, Roca-Oporto C, Rodriguez Pena R, Santos-Perez JL, Rodriguez-Gallego C, Neth O. Executive Summary of the Consensus Document on the Diagnosis and Management of Patients with Primary Immunodeficiencies. Enferm Infecc Microbiol Clin (Engl Ed). 2020 Nov;38(9):438-443. doi: 10.1016/j.eimc.2020.07.001. English, Spanish. PMID 33161954
- [Background] Bierry G, Boileau J, Barnig C, Gasser B, Korganow AS, Buy X, Jeung MY, Roy C, Gangi A. Thoracic manifestations of primary humoral immunodeficiency: a comprehensive review. Radiographics. 2009 Nov;29(7):1909-20. doi: 10.1148/rg.297095717. PMID 19926753
- [Background] Herriot R, Sewell WA. Antibody deficiency. J Clin Pathol. 2008 Sep;61(9):994-1000. doi: 10.1136/jcp.2007.051177. PMID 18755724
- [Background] BRUTON OC. Agammaglobulinemia. Pediatrics. 1952 Jun;9(6):722-8. No abstract available. PMID 14929630
- [Background] Hartung HP, Mouthon L, Ahmed R, Jordan S, Laupland KB, Jolles S. Clinical applications of intravenous immunoglobulins (IVIg)--beyond immunodeficiencies and neurology. Clin Exp Immunol. 2009 Dec;158 Suppl 1(Suppl 1):23-33. doi: 10.1111/j.1365-2249.2009.04024.x. PMID 19883421
- [Background] Hoffmann F, Grimbacher B, Thiel J, Peter HH, Belohradsky BH; Vivaglobin Study Group. Home-based subcutaneous immunoglobulin G replacement therapy under real-life conditions in children and adults with antibody deficiency. Eur J Med Res. 2010 Jun 28;15(6):238-45. doi: 10.1186/2047-783x-15-6-238. PMID 20696632
- [Background] World Health Organization (2005) Recommendations for the production, control and regulation of human plasma for fractionation, Annex 4, TRS nº 941, pp. 69.
- [Background] Radosevich M, Burnouf T. Intravenous immunoglobulin G: trends in production methods, quality control and quality assurance. Vox Sang. 2010 Jan;98(1):12-28. doi: 10.1111/j.1423-0410.2009.01226.x. Epub 2009 Jul 29. PMID 19660029
- [Background] Blasczyk R, Westhoff U, Grosse-Wilde H. Soluble CD4, CD8, and HLA molecules in commercial immunoglobulin preparations. Lancet. 1993 Mar 27;341(8848):789-90. doi: 10.1016/0140-6736(93)90563-v. PMID 8096001
- [Background] Mouthon L, Kaveri SV, Spalter SH, Lacroix-Desmazes S, Lefranc C, Desai R, Kazatchkine MD. Mechanisms of action of intravenous immune globulin in immune-mediated diseases. Clin Exp Immunol. 1996 May;104 Suppl 1:3-9. PMID 8625540
- [Background] Orange JS, Hossny EM, Weiler CR, Ballow M, Berger M, Bonilla FA, Buckley R, Chinen J, El-Gamal Y, Mazer BD, Nelson RP Jr, Patel DD, Secord E, Sorensen RU, Wasserman RL, Cunningham-Rundles C; Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. Use of intravenous immunoglobulin in human disease: a review of evidence by members of the Primary Immunodeficiency Committee of the American Academy of Allergy, Asthma and Immunology. J Allergy Clin Immunol. 2006 Apr;117(4 Suppl):S525-53. doi: 10.1016/j.jaci.2006.01.015. PMID 16580469
- [Background] Bonilla FA, Barlan I, Chapel H, Costa-Carvalho BT, Cunningham-Rundles C, de la Morena MT, Espinosa-Rosales FJ, Hammarstrom L, Nonoyama S, Quinti I, Routes JM, Tang ML, Warnatz K. International Consensus Document (ICON): Common Variable Immunodeficiency Disorders. J Allergy Clin Immunol Pract. 2016 Jan-Feb;4(1):38-59. doi: 10.1016/j.jaip.2015.07.025. Epub 2015 Nov 7. PMID 26563668
- [Background] Yazdani R, Habibi S, Sharifi L, Azizi G, Abolhassani H, Olbrich P, Aghamohammadi A. Common Variable Immunodeficiency: Epidemiology, Pathogenesis, Clinical Manifestations, Diagnosis, Classification, and Management. J Investig Allergol Clin Immunol. 2020;30(1):14-34. doi: 10.18176/jiaci.0388. Epub 2019 Feb 11. PMID 30741636
- [Background] Busse PJ, Razvi S, Cunningham-Rundles C. Efficacy of intravenous immunoglobulin in the prevention of pneumonia in patients with common variable immunodeficiency. J Allergy Clin Immunol. 2002 Jun;109(6):1001-4. doi: 10.1067/mai.2002.124999. PMID 12063531
- [Background] Pourpak Z, Aghamohammadi A, Sedighipour L, Farhoudi A, Movahedi M, Gharagozlou M, Chavoshzadeh Z, Jadid L, Rezaei N, Moin M. Effect of regular intravenous immunoglobulin therapy on prevention of pneumonia in patients with common variable immunodeficiency. J Microbiol Immunol Infect. 2006 Apr;39(2):114-20. PMID 16604243
- [Background] Salehzadeh M, Aghamohammadi A, Rezaei N. Evaluation of immunoglobulin levels and infection rate in patients with common variable immunodeficiency after immunoglobulin replacement therapy. J Microbiol Immunol Infect. 2010 Feb;43(1):11-7. doi: 10.1016/S1684-1182(10)60002-3. Epub 2010 Mar 29. PMID 20434118
- [Background] Suri D, Rawat A, Singh S. X-linked Agammaglobulinemia. Indian J Pediatr. 2016 Apr;83(4):331-7. doi: 10.1007/s12098-015-2024-8. Epub 2016 Feb 24. PMID 26909497
- [Background] Milito C, Pulvirenti F, Pesce AM, Digiulio MA, Pandolfi F, Visentini M, Quinti I. Adequate patient's outcome achieved with short immunoglobulin replacement intervals in severe antibody deficiencies. J Clin Immunol. 2014 Oct;34(7):813-9. doi: 10.1007/s10875-014-0081-9. Epub 2014 Jul 22. PMID 25047154
- [Background] Quinti I, Soresina A, Guerra A, Rondelli R, Spadaro G, Agostini C, Milito C, Trombetta AC, Visentini M, Martini H, Plebani A, Fiorilli M; IPINet Investigators. Effectiveness of immunoglobulin replacement therapy on clinical outcome in patients with primary antibody deficiencies: results from a multicenter prospective cohort study. J Clin Immunol. 2011 Jun;31(3):315-22. doi: 10.1007/s10875-011-9511-0. Epub 2011 Mar 2. PMID 21365217
- [Background] Primary immunodeficiency diseases. Report of an IUIS Scientific Committee. International Union of Immunological Societies. Clin Exp Immunol. 1999 Oct;118 Suppl 1(Suppl 1):1-28. doi: 10.1046/j.1365-2249.1999.00109.x. No abstract available. PMID 10540200
- [Background] EMA/CHMP/BPWP/94033/2007 rev. 4. Guideline on the clinical investigation of human normal immunoglobulin for intravenous administration (IVIg), Sep,2020.
- [Background] Guidance for Industry: Safety, Efficacy, and Pharmacokinetic Studies to Support Marketing of Immune Globulin Intravenous (Human) as Replacement Therapy for Primary Humoral Immunodeficiency. Rockville, MD, pp. 17, Jun,2008.
- [Background] Brasil, Resolução nº 251, de 07 de agosto de 1977. Disponível em; https://www.inca.gov.br/sites/ufu.sti.inca.local/files//media/document//resolucao-cns-251-97.pdf. Acesso em 25 de out de 2023
- [Background] Mongkonsritragoon W, Srivastava R, Seth D, Navalpakam A, Poowuttikul P. Non-infectious Pulmonary Complications in Children with Primary Immunodeficiency. Clin Med Insights Pediatr. 2023 Sep 8;17:11795565231196431. doi: 10.1177/11795565231196431. eCollection 2023. PMID 37692068
- [Background] World Health Organization (2009). Conceptual Framework of the International Classification for Patient safety. World Health Organization, Patient Safety. Quem Press.
- [Background] Brasil. Manual de orientação: pendências frequentes em protocolo de pesquisas. Disponível em: https://conselho.saude.gov.br/Web_comissoes/conep/aquivos/documentos/MANUAL_ORIENTACAO_PENDENCIAS_FREQUENTES_PROTOCOLOS_PESQUISA_CLINICA_V1.pdf. Acesso em: 26out2023
- [Background] Harmonisation for better health (1998). Statitical Principles for Clinical Trials E9. Disponível em: Disponível em: https://database.ich.org/sites/default/files/E9_Guideline.pdf Acesso em: 01nov2023
- [Background] Harmonisation for better health (1998). The Guideline Statistical Principles for Clinical Trials E9 (R1). Disponível em: https://database.ich.org/sites/default/files/E9-R1_Step4_Guideline_2019_1203.pdf Acesso em: 01nov2023
- [Background] Conselho das Organizações Internacionais de Ciências Médicas (CIOMS) em colaboração com a Organização Mundial da Saúde (2016). Diretrizes éticas internacionais para pesquisas relacionadas a saúde envolvendo seres humanos. Disponível em: https://cioms.ch/wp-content/uploads/2018/11/CIOMS-final-Diretrizes-Eticas-Internacionais-Out18.pdf. Acesso em: 31out2023
- [Background] Harmonisation for better health (2016). Guideline for Good Clinical Practice. Disponível em: https://database.ich.org/sites/default/files/E6_R2_Addendum.pdf Acesso em: 01nov2023
- [Background] Organização Pan-Americana da Saúde (2005). Boas Práticas Clínicas: Documentos das Américas. Disponível em: https://www.gov.br/anvisa/ptbr/centraisdeconteudo/publicacoes/medicamentos/pesquisa-clinica/manuais-e-guias/documento-das-americas-boas-praticas-clinicas.pdf/view. Acesso em: 01out2023
- [Background] Brasil (2018). Lei Geral de Proteção de Dados. 14ago2018. Disponível em: https://www.planalto.gov.br/ccivil_03/_ato2015-2018/2018/lei/L13709compilado.htm. Acessado em 09nov23.
- [Background] Brasil (2008) Diretrizes Operacionais para o estabelecimento e o funcionamento de comitês de monitoramento de dados e segurança. Brasília, pp. 44.
- [Background] Food and Drug Administration (2006). Guidance for Clinical Trial Sponsors on the Establishment and Operation of Clinical Trial Data Monitoring Committees. Rockville, MD, pp. 38.